CLINICAL TRIAL: NCT04166526
Title: A Pilot Study on Neuroimaging in SCD: Part of The Boston Consortium to Cure Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ellen Grant, Director, FNNDSC, Boston Children's Hospital
Other Study IDs: IRB-P00033322; 1OT2HL152640-01 (NIH)
Record Dates: First submitted 2019-10-15; First posted 2019-11-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell; MRI; Near Infrared Spectroscopy (NIRS)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Typically developing children: Participants of this group will not have a diagnosis of SCD. These participants will undergo an MRI, lasting approximately an hour, with simultaneous FDNIRS-DCS monitoring.
  Interventions: Device: FDNIRS-DCS; Device: MRI
- Group 2: Children with SCD not receiving treatment: Participants of this group have a diagnosis of SCD, but do not receive chronic transfusions, gene therapy or bone marrow transplants. These participants will undergo an MRI, lasting approximately an hour, with simultaneous FDNIRS-DCS monitoring.
  Interventions: Device: FDNIRS-DCS; Device: MRI
- Group 3: Children with SCD who have undergone gene therapy: Participants of this group have a diagnosis of SCD and have had gene therapy at least one month prior to enrollment. These participants will undergo an MRI, lasting approximately an hour, with simultaneous FDNIRS-DCS monitoring.
  Interventions: Device: FDNIRS-DCS; Device: MRI
- Group 4: Children with SCD who have chronic transfusions: Participants of this group have a diagnosis of SCD and receive chronic transfusions. These participants will undergo an MRI, lasting approximately an hour, with simultaneous FDNIRS-DCS monitoring.
  Interventions: Device: FDNIRS-DCS; Device: MRI

INTERVENTIONS:
Device: FDNIRS-DCS — FDNIRS-DCS measurements will be performed at the same time as all MRI scans. Participants in Group 4 will have additional measurements before, during, and after the their scheduled transfusion.
  Other Names: Frequency-Domain Near-Infrared and Diffuse Correlation Spectroscopy
Device: MRI — Participants in Groups 1-3 will receive a single, hour-long MRI. Participants in Group 4 will receive two, one hour long MRI scans: one within a week prior to their transfusion and one within a week after their transfusion.
  Other Names: Magnetic Resonance Imaging

SUMMARY:
Sickle Cell Disease (SCD) impairs oxygen transport to tissue and causes endothelial injury. Thus, therapeutic interventions aim to improve both, but there is an unmet need for biomarkers to determine when intervention is necessary and evaluate the effectiveness of the chosen intervention in individual patients. This study proposes to monitor SCD and its treatment through their impact on cerebral hemodynamics, as the brain is one of the most vulnerable and consequential targets of the disease. Specifically, this study will optimize quantitative magnetic resonance imaging (MRI) and advanced optical spectroscopy techniques such as frequency-domain near-infrared and diffuse correlation spectroscopies (FDNIRS-DCS) to monitor 1) cerebral oxygen transport with measures of cerebral blood flow (CBF), cerebral oxygen extraction fraction (OEF) and cerebral metabolic rate of oxygen consumption (CMRO2) and 2) endothelial function with cerebrovascular reactivity (CVR).

Additionally, this study aims to monitor baseline cerebral oxygen transport and CVR, as well as changes that occur with treatment (transfusion or genetic therapy to induce fetal hemoglobin) and assess hemoglobinopathy patients with known genotypes and phenotypes. The ultimate goal is to demonstrate the potential of this monitoring approach to select individual SCD subjects for interventions and evaluate individual responses to treatment. Success will help justify inclusion of these modalities in ongoing and future clinical trials of novel SCD therapies.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (healthy controls):

* Children ages 8-18 without SCD

Group 2 (SCD patients without treatment):

* SCD patients ages 8-18 who:

  * have not undergone gene therapy or a bone marrow transplant
  * are not receiving chronic transfusions
  * have not received a blood transfusion in the past 3 months

Group 3 (SCD patients who have undergone gene therapy):

* SCD patients ages 8-18 who have had gene therapy at least one month prior to enrollment

Group 4 (SCD patients who have chronic transfusions):

* SCD patients ages 8-18 who receive chronic transfusions

Exclusion Criteria:

* Electrical implants such as cardiac pacemakers or perfusion pumps;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prosthesis, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants;
* Ferromagnetic objects such as jewelry or metal clips;
* Women of childbearing age who are seeking to become pregnant, who are breastfeeding, or who suspect they may be pregnant;
* Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions;
* Any greater than normal potential for cardiac arrest;
* Subjects requiring sedation for MRI

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In this pilot study, investigators plan on recruiting 8 children between the ages of 8-18 from hematology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of FDNIRS-DCS in measuring blood oxygenation of the brain | 6 months
  Blood oxygenation of the brain will be measured using FDNIRS-DCS techniques and then compared with data from a simultaneous MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Grant, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No